CLINICAL TRIAL: NCT04071496
Title: Development of an Approach for the Differential Diagnosis of Chronic Idiopathic Thrombocytopenic Purpura and Congenital Thrombocytopenia
Brief Title: Diagnostic of Chronic Thrombocytopenia
Acronym: DIATROC
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2008/06
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Congenital Thrombocytopenia; Chronic Idiopathic Thrombocytopenic Purpura
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 dry tube of 5 ml, 3 citrated tubes of 5 ml, 1 tube citrate dextrose acid of 7 ml
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood samples — 1 dry tube of 5 ml, 3 citrated tubes of 5 ml, 1 tube citrate dextrose acid of 7 ml

SUMMARY:
The objective of this study is to provide simple and relevant clinical and biological elements to distinguish a possible Congenital Thrombocytopenia from a Chronic Idiopathic Thrombocytopenic Purpura .

DETAILED DESCRIPTION:
Congenital Thrombocytopenia is a group of rare diseases, often unrecognized and misdiagnosed as Chronic Idiopathic Thrombocytopenic Purpura. These Chronic Idiopathic Thrombocytopenic Purpura, which are exclusion diagnoses, are most often treated with corticosteroids or intravenous immunoglobulins and sometimes, when thrombocytopenia is refractory, splenectomy is performed. Currently, it is often before a case of thrombocytopenia refractory to the treatment of the dysimmunity syndrome that the notion of Congenital Thrombocytopenia is evoked. The percentage of false diagnoses (misdiagnosed Chronic Idiopathic Thrombocytopenic Purpura diagnoses) seems to represent to date 10 to 20% of cases.

The objective of this study is to provide simple and relevant clinical and biological elements to distinguish a possible Congenital Thrombocytopenia from a Chronic Idiopathic Thrombocytopenic Purpura.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic thrombocytopenia (> 6 months) between 10 and 150 G / L, regardless of age or gender,
* Subjects with a definite Chronic Idiopathic thrombocytopenic purpuras, - Subjects with a certain degree of certainty, sometimes pre-identified and already known at the level of the C reactive protein,
* Subjects with chronic thrombocytopenia of undetermined origin, not definitively entering one of the 2 groups mentioned above.

Exclusion Criteria:

* Thrombocytopenia less than 6 months old;
* Patients with thrombocytopenia related to a viral or chronic infectious pathology (HIV infections or hepatitis C virus, bacterial infections with Helicobacter pillory, for example), an autoimmune disease, in particular systemic lupus and / or antiphospholipid syndrome, a bleeding disorder such as a Intra-vascular Disseminated coagulation, thrombotic microangiopathy, hypersplenism, a responsible medication intake, myelodysplastic syndrome, a pregnancy in progress.
* Patients should not be treated with Immunoglobulin IV, rituximab or anti-CD20 less than 30 days before the date of collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Congenital Thrombocytopenia Patients and Chronic Idiopathic Thrombocytopenic Purpura Patients
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-11-25 (Actual); Primary Completion 2012-03-12 (Actual); Study Completion 2012-03-12 (Actual)

PRIMARY OUTCOMES:
Modelization of congenital thrombocytopenia test | AT the screening
  Taking into account the clinical and biological data of patients (flow cytometry and electron microscopy), validation using resampling methods (bootstrap, jacknife, cross validation ...)
Modelization of chronic idiopathic thrombocytopenic purpura test | AT the screening
  Taking into account the clinical and biological data of patients (flow cytometry and electron microscopy), validation using resampling methods (bootstrap, jacknife, cross validation ...)

CONTACTS AND LOCATIONS:
Overall Officials: Paquita NURDEN, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No